CLINICAL TRIAL: NCT01617096
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Phase 3 Safety and Effectiveness Trial of a Vaginal Matrix Ring Containing Dapivirine for the Prevention of HIV-1 Infection in Women
Brief Title: Phase 3 Safety and Effectiveness Trial of Dapivirine Vaginal Ring for Prevention of HIV-1 in Women
Acronym: ASPIRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MTN-020; UM1AI068633-06 (NIH)
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Results first posted 2022-12-16 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: HIV Infections
Keywords: HIV Infections; Anti-HIV agents; HIV-1
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dapivirine Vaginal Ring (Experimental): Vaginal ring containing 25mg dapivirine
  Interventions: Combination Product: Dapivirine Vaginal Ring
- Placebo Ring (Placebo Comparator): Vaginal ring containing no drug substance
  Interventions: Combination Product: Placebo Ring

INTERVENTIONS:
Combination Product: Dapivirine Vaginal Ring — Dosage form: vaginal ring Dosage: 25mg Frequency: monthly Duration: 12 months
  Arms: Dapivirine Vaginal Ring
Combination Product: Placebo Ring — Vaginal ring containing no drug substance
  Arms: Placebo Ring

SUMMARY:
This is a double-blind, randomised, placebo-controlled study to assess the safety and efficacy of a silicone elastomer vaginal matrix ring.

DETAILED DESCRIPTION:
A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Phase 3 Safety and Effectiveness Trial of a Vaginal Matrix Ring Containing Dapivirine for the Prevention of HIV-1 Infection in Women." MTN-020 will enroll approximately 3676 sexually active HIVnegative women aged 18-45 years randomized in a 1:1 ratio to receive either a vaginal ring containing 25 mg of dapivirine or a placebo vaginal ring. Rings will be inserted once every 28 days for 12 consecutive months. MTN expects to initiate this study in August 2012.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 45 years (inclusive) at screening, verified per site SOPs; within this range, sites may restrict the upper age limit per site SOPs, to target women at high risk of HIV infection
* Able and willing to provide written informed consent to be screened for and to take part in the study
* Able and willing to provide adequate locator information, as defined in site SOPs
* HIV-uninfected based on testing performed by study staff at screening and enrollment (per applicable algorithm in Appendix II)
* Per participant report, sexually active, defined as having vaginal intercourse at least once in the 3 months prior to screening
* Using an effective method of contraception at enrollment, and intending to use an effective method for the duration of study participation; effective methods include hormonal methods (except contraceptive ring); intrauterine device (IUD); and sterilization (of participant, as defined in site SOPs)
* At screening and enrollment, agrees not to participate in other research studies involving drugs, medical devices, vaginal products, or vaccines for the duration of study participation -- Note: Tampons may be used for the duration of the trial.

Exclusion Criteria:

* Per participant report at screening:

  * Intends to become pregnant during study participation
  * Plans to relocate away from the study site during study participation
  * Plans to travel away from the study site for more than 8 consecutive weeks during study participation
* Is pregnant

  -- Note: A documented negative pregnancy test performed by study staff is required for inclusion; however a self-reported pregnancy is adequate for exclusion from the study.
* Currently breastfeeding
* Diagnosed with urinary tract infection (UTI)

  -- Note: Otherwise eligible participants diagnosed with UTI during screening are offered treatment and may be enrolled after completing treatment and all symptoms have resolved. If treatment is completed and symptoms have resolved within 28 days of obtaining informed consent for screening, the participant may be enrolled.
* Diagnosed with pelvic inflammatory disease, an STI or reproductive tract infection (RTI) requiring treatment per current WHO guidelines

  -- Note: Otherwise eligible participants diagnosed during screening with pelvic inflammatory disease or STI/RTI requiring treatment per WHO guidelines - other than asymptomatic BV and asymptomatic candidiasis - are offered treatment and may be enrolled after completing treatment and all symptoms have resolved. If treatment is completed and symptoms have resolved within 28 days of obtaining informed consent for screening, the participant may be enrolled. Genital warts requiring treatment also must be treated prior to enrollment. Genital warts requiring therapy are defined as those that cause undue burden or discomfort to the participant, including bulky size, unacceptable appearance, or physical discomfort.
* Has a clinically apparent Grade 2 or higher pelvic exam finding (observed by study staff) as per the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 1.0, December, 2004 (Clarification dated August 2009), Addendum 1-Female Genital Grading Table for Use in Microbicide Studies

  * Note: Cervical bleeding associated with speculum insertion and/or specimen collection judged to be within the range of normal according to the clinical judgment of the Investigator of Record (IoR)/designee is considered expected non-menstrual bleeding and is not exclusionary.
  * Note: Otherwise eligible participants with exclusionary pelvic exam findings may be enrolled/randomized after the findings have improved to a non-exclusionary severity grading or resolved. If improvement to a non-exclusionary grade or resolution is documented within 28 days of providing informed consent for screening, the participant may be enrolled.
* Participant report and/or clinical evidence of any of the following:

  * Known adverse reaction to any of the study products (ever)
  * Known adverse reaction to latex (ever)
  * Chronic vaginal candidiasis
  * Non-therapeutic injection drug use in the 12 months prior to Screening
  * Post-exposure prophylaxis (PEP) for HIV exposure within 6 months prior to enrollment
  * Last pregnancy outcome 90 days or less prior to enrollment
  * Gynecologic or genital procedure (e.g., tubal ligation, dilation and curettage, piercing) 90 days or less prior to enrollment
  * Recent participation in any other research study involving drugs, medical devices, vaginal products, or vaccines, within 60 days of enrollment
  * Participation in the MTN-003, Vaginal and Oral Interventions to Control the Epidemic (VOICE) clinical trial, or any other HIV prevention study using systemic or topical antiretroviral medications, within 12 months of enrollment
  * As determined by the IoR/designee, any significant uncontrolled active or chronic cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, endocrine, respiratory, immunologic disorder or infectious disease, including active tuberculosis
* Has any of the following laboratory abnormalities at Screening Visit:

  * Aspartate aminotransferase (AST) or alanine transaminase (ALT) Grade 1 or higher as per the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 1.0, December, 2004 (Clarification dated August 2009)
  * Creatinine Grade 2 or higher as per the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 1.0, December, 2004 (Clarification dated August 2009)
  * Hemoglobin Grade 2 or higher as per the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 1.0, December, 2004 (Clarification dated August 2009)
  * Platelet count Grade 1 or higher as per the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 1.0, December, 2004 (Clarification dated August 2009)
  * Pap result Grade 2 or higher according to the Female Genital Grading Table for Use in Microbicide Studies Addendum 1 to the DAIDS Table for Grading Adult and Pediatric Adverse Events, Version 1.0, December 2004 (Clarification dated August 2009)

    * Note: Otherwise eligible participants with an exclusionary test may be re-tested during the screening process.
    * Note: Women with a documented normal result within the 12 months prior to enrollment need not have Pap smear during the screening period. Women with a Grade 1 abnormal Pap smear can be enrolled upon completion of the initial phase of evaluation if no current treatment is indicated (based on local standard of care for management of abnormal cervical cytology). Need for a repeat Pap within 6 months does not preclude enrollment prior to that result becoming available.
* Has any other condition that, in the opinion of the IoR/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2629 (Actual)
Dates: Start 2012-07-24 (Actual); Primary Completion 2015-07-03 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jared Baeten, MD, PhD, Study Chair — International Clinical Research Center, Department of Global Health, University of Washington; Thesla Palanee, PhD, Study Chair — Wits Reproductive Health and HIV Institute (WRHI), Research Centre
Locations (7):
- Malawi (2):
  - College of Medicine - Johns Hopkins University Research Project, Blantyre
  - UNC Project, Lilongwe
- South Africa (3):
  - CAPRISA, eThekwini Clinical Research Site, Durban, KwaZulu-Natal
  - Desomond Tutu HIV Center, Cape Town
  - Wits Reproductive Health and HIV Institute, Johannesburg
- MU-JHU Care LTD, MU-JHU Research Collaboration, Kampala, Uganda
- UZ-Obstetrics & Gynecology Research Clinic at Spillhaus, Belgravia, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stalter RM, Dong TQ, Hendrix CW, Palanee-Phillips T, van der Straten A, Hillier SL, Kiweewa FM, Mgodi NM, Marzinke MA, Bekker LG, Soto-Torres L, Baeten JM, Brown ER; MTN-020/ASPIRE Study Team. Assessing Per-Sex-Act HIV-1 Risk Reduction Among Women Using the Dapivirine Vaginal Ring. J Infect Dis. 2024 Apr 12;229(4):1158-1165. doi: 10.1093/infdis/jiad550. PMID 38099506
- [Derived] Browne EN, Brown ER, Palanee-Phillips T, Reddy K, Naidoo L, Jeenarain N, Nair G, Husnik MJ, Singh D, Scheckter R, Soto-Torres L, Baeten JM, van der Straten A; MTN-020/ASPIRE Study Team. Patterns of Adherence to a Dapivirine Vaginal Ring for HIV-1 Prevention Among South African Women in a Phase III Randomized Controlled Trial. J Acquir Immune Defic Syndr. 2022 Aug 1;90(4):418-424. doi: 10.1097/QAI.0000000000002990. PMID 35344520
- [Derived] Leslie J, Kiweewa F, Palanee-Phillips T, Bunge K, Mhlanga F, Kamira B, Baeten J, Katz A, Hillier S, Montgomery E; MTN-020/ASPIRE Study Team. Experiences with simultaneous use of contraception and the vaginal ring for HIV prevention in sub-Saharan Africa. BMC Womens Health. 2021 Apr 23;21(1):175. doi: 10.1186/s12905-021-01321-5. PMID 33892693
- [Derived] Mayo AJ, Browne EN, Montgomery ET, Torjesen K, Palanee-Phillips T, Jeenarain N, Seyama L, Woeber K, Harkoo I, Reddy K, Tembo T, Mutero P, Tauya T, Chitukuta M, Gati Mirembe B, Soto-Torres L, Brown ER, Baeten JM, van der Straten A; MTN-020/ASPIRE study team. Acceptability of the Dapivirine Vaginal Ring for HIV-1 Prevention and Association with Adherence in a Phase III Trial. AIDS Behav. 2021 Aug;25(8):2430-2440. doi: 10.1007/s10461-021-03205-z. Epub 2021 Mar 13. PMID 33713213
- [Derived] Palanee-Phillips T, Brown ER, Szydlo D, Matovu Kiweewa F, Pather A, Harkoo I, Nair G, Soto-Torres L, Hillier SL, Baeten JM; MTN-020/ASPIRE Study Team. Risk of HIV-1 acquisition among South African women using a variety of contraceptive methods in a prospective study. AIDS. 2019 Aug 1;33(10):1619-1622. doi: 10.1097/QAD.0000000000002260. PMID 31306167
- [Derived] Kiweewa FM, Brown E, Mishra A, Nair G, Palanee-Phillips T, Mgodi N, Nakabiito C, Chakhtoura N, Hillier SL, Baeten JM; MTN-020/ASPIRE Study Team. Acquisition of Sexually Transmitted Infections among Women Using a Variety of Contraceptive Options: A prospective Study among High-risk African Women. J Int AIDS Soc. 2019 Feb;22(2):e25257. doi: 10.1002/jia2.25257. PMID 30816632
- [Derived] Riddler SA, Balkus JE, Parikh UM, Mellors JW, Akello C, Dadabhai S, Mhlanga F, Ramjee G, Mayo AJ, Livant E, Heaps AL, O'Rourke C, Baeten JM; MTN-015 and MTN-020/ASPIRE Study Teams. Clinical and Virologic Outcomes Following Initiation of Antiretroviral Therapy Among Seroconverters in the Microbicide Trials Network-020 Phase III Trial of the Dapivirine Vaginal Ring. Clin Infect Dis. 2019 Jul 18;69(3):523-529. doi: 10.1093/cid/ciy909. PMID 30346511
- [Derived] Mensch BS, Richardson BA, Husnik M, Brown ER, Kiweewa FM, Mayo AJ, Baeten JM, Palanee-Phillips T, van der Straten A; MTN-020/ASPIRE study team. Vaginal Ring Use in a Phase 3 Microbicide Trial: A Comparison of Objective Measures and Self-reports of Non-adherence in ASPIRE. AIDS Behav. 2019 Feb;23(2):504-512. doi: 10.1007/s10461-018-2261-8. PMID 30218318
- [Derived] Baeten JM, Palanee-Phillips T, Brown ER, Schwartz K, Soto-Torres LE, Govender V, Mgodi NM, Matovu Kiweewa F, Nair G, Mhlanga F, Siva S, Bekker LG, Jeenarain N, Gaffoor Z, Martinson F, Makanani B, Pather A, Naidoo L, Husnik M, Richardson BA, Parikh UM, Mellors JW, Marzinke MA, Hendrix CW, van der Straten A, Ramjee G, Chirenje ZM, Nakabiito C, Taha TE, Jones J, Mayo A, Scheckter R, Berthiaume J, Livant E, Jacobson C, Ndase P, White R, Patterson K, Germuga D, Galaska B, Bunge K, Singh D, Szydlo DW, Montgomery ET, Mensch BS, Torjesen K, Grossman CI, Chakhtoura N, Nel A, Rosenberg Z, McGowan I, Hillier S; MTN-020-ASPIRE Study Team. Use of a Vaginal Ring Containing Dapivirine for HIV-1 Prevention in Women. N Engl J Med. 2016 Dec 1;375(22):2121-2132. doi: 10.1056/NEJMoa1506110. Epub 2016 Feb 22. PMID 26900902

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants provided written informed consent were invited to screen for the clinical trial. Each participant engaged in the screening process for up to 4 weeks (28 days) prior to enrollment. Participants who complied with inclusion and exclusion criteria were invited to enroll in the trial. Participants were randomized in a 1:1 ratio to either the Dapivirine Vaginal Ring or placebo ring group.
Pre-assignment Details: Healthy, sexually active HIV-negative women who provided written informed consent were invited to screen for the clinical trial. Each participant engaged in the screening process for up to 4 weeks (28 days) prior to enrollment. Participants who complied with all the inclusion and none of the exclusion criteria were invited to enroll in the clinical trial. Eligible participants were randomly assigned in a 1:1 ratio to either the Dapivirine Vaginal Ring-004 or placebo ring group.
Period: Overall Study
Arm/Group | Dapivirine Vaginal Ring | Placebo Ring
Started | 1313 | 1316
Completed | 1165 | 1179
Not Completed | 148 | 137
Not completed — Withdrawal by Subject | 96 | 81
Not completed — Lost to Follow-up | 37 | 32
Not completed — Physician Decision | 10 | 18
Not completed — Death | 4 | 3
Not completed — Other | 1 | 3

BASELINE CHARACTERISTICS:
Population: Primary safety cohort
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapivirine Vaginal Ring | Placebo Ring | Total
Number analyzed (Participants) | 1313 | 1316 | 2629
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.2 (6.09) | 27.3 (6.28) | 27.2 (6.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1313 | 1316 | 2629
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 3 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1228 | 1226 | 2454
  White | 2 | 0 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 70 | 87 | 157
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 713 | 713 | 1426
  Zimbabwe | 338 | 340 | 678
  Malawi | 135 | 137 | 272
  Uganda | 127 | 126 | 253
BMI [Mean (Standard Deviation); unit: kg/(m^2)] | 26.8 (6.41) | 27.2 (6.93) | 27.0 (6.68)
Education Status [Count of Participants; unit: Participants]
  Less than Secondary School | 212 | 192 | 404
  Secondary School and Higher | 1101 | 1124 | 2225
Marital Status [Count of Participants; unit: Participants]
  Married | 527 | 547 | 1074
  Non-Married | 786 | 767 | 1553
  Missing | 0 | 2 | 2
Has children [Count of Participants; unit: Participants] | 1188 | 1177 | 2365
Has main partner [Count of Participants; unit: Participants]
  Yes | 1307 | 1309 | 2616
  Missing | 0 | 1 | 1
  No | 6 | 6 | 12
Presence of STIs [Count of Participants; unit: Participants] | 268 | 265 | 533
Partner knowledge of ring use [Count of Participants; unit: Participants]
  Yes | 835 | 845 | 1680
  Missing | 0 | 1 | 1
  No | 478 | 470 | 948
Number of sex partners in the last 3 months [Count of Participants; unit: Participants]
  0-1 partners | 1101 | 1089 | 2190
  >2 | 212 | 227 | 439

OUTCOME MEASURES:

1. Primary Outcome: Efficacy as Determined by the Proportion of Women in Each Arm With HIV-1 Seroconversion After 120 Endpoints Are Observed in the Trial.
Description: The primary endpoint is HIV-1 seroconversion as measured by rapid and specialised laboratory testing according to comprehensive HIV testing algorithm. Endpoint confirmation of HIV infection is by Western Blot.
Time Frame: minimum of 12 months and a maximum of 14 months per participant
Population: The primary effectiveness Cohort included all eligible randomised participants excluding participants deemed to be HIV-1 RNA positive at the time of randomization, based on retrospective PCR testing of stored blood samples taken at enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapivirine Vaginal Ring | Placebo Ring
Number analyzed (Participants) | 1313 | 1313
Participants | 71 | 97

2. Primary Outcome: The Number of Participants That Experienced Grade 2, 3, 4 and Serious Adverse Events Over the Investigational Product Used Period (25 mg Dapivirine Administered in a Silicone Elastomer Vaginal Matrix Ring (DVR), Inserted Once Every 4 Weeks).
Description: Participants with grade 2 adverse events, judged to be related to investigational product, grade 3 and grade 4 adverse events and all serious adverse events.
  DAIDS severity grades are defined as follows:
  Grade 1 = mild Grade 2 = moderate Grade 3 = severe Grade 4 = potentially life-threatening Grade 5 = death
Time Frame: minimum of 12 months and a maximum of 14 months per participant
Population: The Primary Safety Cohort (or ITT Cohort) included all eligible, randomized participants. All participants were analyzed as members of the treatment group to which they were randomized regardless of adherence to the planned course of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapivirine Vaginal Ring | Placebo Ring
Number analyzed (Participants) | 1313 | 1316
Participants | 1237 | 1231

3. Secondary Outcome: Adherence to the Dapivirine Vaginal Ring.
Description: Dapivirine residual levels in used rings and dapivirine plasma concentrations are two objective measures of adherence to DVR ring use.
  Adherence was defined as a dapivirine ring residual level <=23.5 mg and dapivirine plasma level >= 95 pg/mL.
Time Frame: 12 months per participant
Population: Adherence is defined by a dapivirine residual level in returned used rings ≤ 23.5 mg and a dapivirine plasma concentration ≥ 95 pg/mL (if they are both available; otherwise categorisation was based on the available measurement. The objective measures (dapivirine residual levels in used rings and dapivirine plasma concentrations) used can only be determined for participants who used the active vaginal dapivirine ring.
Measure: Number; unit: participants with data
Arm/Group | Dapivirine Vaginal Ring
Number analyzed (Participants) | 1288
participants with data
  Month 1: number analyzed (Participants) | 503
  Month 1 | 443
  Month 2: number analyzed (Participants) | 551
  Month 2 | 460
  Month 3: number analyzed (Participants) | 1281
  Month 3 | 953
  Month 4: number analyzed (Participants) | 645
  Month 4 | 537
  Month 5: number analyzed (Participants) | 675
  Month 5 | 573
  Month 6: number analyzed (Participants) | 1239
  Month 6 | 963
  Month 7: number analyzed (Participants) | 788
  Month 7 | 687
  Month 8: number analyzed (Participants) | 834
  Month 8 | 699
  Month 9: number analyzed (Participants) | 1205
  Month 9 | 943
  Month 10: number analyzed (Participants) | 990
  Month 10 | 830
  Month 11: number analyzed (Participants) | 1106
  Month 11 | 916
  Month 12: number analyzed (Participants) | 1179
  Month 12 | 922
  Month 13: number analyzed (Participants) | 1037
  Month 13 | 872
  Month 14: number analyzed (Participants) | 1034
  Month 14 | 858
  Month 15: number analyzed (Participants) | 1040
  Month 15 | 793
  Month 16: number analyzed (Participants) | 875
  Month 16 | 704
  Month 17: number analyzed (Participants) | 870
  Month 17 | 701
  Month 18: number analyzed (Participants) | 876
  Month 18 | 675
  Month 19: number analyzed (Participants) | 756
  Month 19 | 600
  Month 20: number analyzed (Participants) | 753
  Month 20 | 598
  Month 21: number analyzed (Participants) | 759
  Month 21 | 576
  Month 22: number analyzed (Participants) | 644
  Month 22 | 499
  Month 23: number analyzed (Participants) | 638
  Month 23 | 485
  Month 24: number analyzed (Participants) | 644
  Month 24 | 471
  Month 25: number analyzed (Participants) | 520
  Month 25 | 391
  Month 26: number analyzed (Participants) | 519
  Month 26 | 384
  Month 27: number analyzed (Participants) | 523
  Month 27 | 367
  Month 28: number analyzed (Participants) | 362
  Month 28 | 263
  Month 29: number analyzed (Participants) | 361
  Month 29 | 258
  Month 30: number analyzed (Participants) | 361
  Month 30 | 251
  Month 31: number analyzed (Participants) | 175
  Month 31 | 133
  Month 32: number analyzed (Participants) | 170
  Month 32 | 130
  Month 33: number analyzed (Participants) | 170
  Month 33 | 120
  Month 34: number analyzed (Participants) | 6
  Month 34 | 4

4. Secondary Outcome: Acceptability of the DVR and Placebo Vaginal Ring
Description: Questionnaires and qualitative data regarding the acceptability of use of a vaginal ring inserted once every 4 weeks over the trial period; Percentage of participants with positive response. Response of 'likely' or 'very likely' to the question: 'If in the future a vaginal ring was available that provided some protection against HIV, and it was similar to the one you used in this trial, how likely would you be to keep it inserted in your vagina every day?'
Time Frame: 12 months per participant
Population: The Primary Safety Cohort (or ITT Cohort) included all eligible, randomized participants. Acceptability was reported for participant who provided responses to acceptability questionnaires.
Measure: Number; unit: percentage of participants with data
Arm/Group | Dapivirine Vaginal Ring | Placebo Ring
Number analyzed (Participants) | 1072 | 1062
percentage of participants with data | 95.9 | 96.8

5. Secondary Outcome: Human Immunodeficiency Virus Type 1 Drug Resistance Mutations Among Participants Who Acquired HIV-1 Infection.
Description: The analysis of HIV-1 drug resistance will be primarily descriptive in nature, and will depend on the pattern of resistance mutations observed in the HIV-1 seroconverters. The percentage of HIV-1 seroconverters with at least one HIV-1 drug resistant mutation will be presented overall, and by treatment arm, with corresponding 95% CIs.
Time Frame: minimum of 12 months and a maximum of 14 months per participant
Population: The virology population included all ITT participants with seroconversion, excluding those who never received investigational product, or were retrospectively found to be HIV-1 RNA positive at enrollment (m-ITT) or were HIV-1 infected after discontinuation of ring use. Seroconversions among participants who were continued on open-label DVR-004 were included in the DVR-004 group, independent of initial randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapivirine Vaginal Ring | Placebo Ring
Number analyzed (Participants) | 71 | 97
Participants | 68 | 96

ADVERSE EVENTS:
Time Frame: 24 Months
Description: The analysis of AEs was mainly descriptive in nature. The number and percentage of participants who experienced AEs are presented by Medical Dictionary for Regulatory Activities System Organ Class and preferred term, and by treatment group.
  Separate tabulations were created for AEs of special interest, ie, urogenital AEs and STIs. For this purpose, preferred terms were grouped into categories of interest. Urogenital and gynecological AEs were also analyzed separately.
Arm/Group | Dapivirine Vaginal Ring | Placebo Ring
All-Cause Mortality (participants affected / at risk) | 4/1313 | 3/1316
Serious Adverse Events (participants affected / at risk) | 116/1313 | 130/1316
Other Adverse Events (participants affected / at risk) | 1237/1313 | 1041/1316
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapivirine Vaginal Ring (N=1313) | Placebo Ring (N=1316)
Vaginal Discharge (Reproductive system and breast disorders) | 17 (17) | 20 (21)
Pelvic Pain (Reproductive system and breast disorders) | 15 (17) | 20 (22)
Metrorrhagia (Reproductive system and breast disorders) | 16 (17) | 9 (9)
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 10 (11) | 12 (13)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 9 (9) | 5 (7)
Cervix erythema (Reproductive system and breast disorders) | 6 (6) | 5 (5)
Vaginal odour (Reproductive system and breast disorders) | 3 (3) | 8 (8)
Dyspareunia (Reproductive system and breast disorders) | 4 (4) | 2 (2)
Menorrhagia (Reproductive system and breast disorders) | 3 (3) | 3 (3)
Pelvic discomfort (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Cervical dysplasia (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Uterine Pain (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Cervical discharge (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Cervix haemorrage uterine (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Cervix oedema (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Coital bleeding (Reproductive system and breast disorders) | 1 (1) | 1 (2)
Menometrorrhagia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Vaginal erosion (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Vulvovaginal pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Genital discomfort (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pruritius genital (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine Cervical pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine Cervix ulcer (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulvovaginal rash (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 9 (9)
Alanine aminotransferase increased (Investigations) | 3 (3) | 7 (7)
Neutrophil count decreased (Investigations) | 4 (4) | 6 (6)
Haemoglobin decreased (Investigations) | 3 (3) | 1 (1)
White blood cell count decreased (Investigations) | 1 (2) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Cervicitis (Infections and infestations) | 2 (3) | 6 (7)
Vulvovaginitis (Infections and infestations) | 2 (2) | 5 (5)
Urinary tract infection (Infections and infestations) | 2 (2) | 5 (5)
Vulvovaginal candidiasis (Infections and infestations) | 2 (2) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 1 (1)
Application site discomfort (General disorders) | 4 (4) | 2 (2)
Application site pain (General disorders) | 1 (1) | 4 (4)
Suprapubic pain (General disorders) | 0 (0) | 1 (1)
Pollakiurua (Renal and urinary disorders) | 4 (4) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Bladder pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Strangury (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal laceration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dapivirine Vaginal Ring (N=1313) | Placebo Ring (N=1316)
Metrorrhagia (Reproductive system and breast disorders) | 723 | 732
Menorrhagia (Reproductive system and breast disorders) | 259 | 242
Vaginal discharge (Reproductive system and breast disorders) | 179 | 174
Menometrorrhagia (Reproductive system and breast disorders) | 160 | 148
Vulvovaginal pruritus (Reproductive system and breast disorders) | 128 | 135
Cervical dysplasia (Reproductive system and breast disorders) | 127 | 123
Pelvic pain (Reproductive system and breast disorders) | 42 | 46
Vulval ulceration (Reproductive system and breast disorders) | 29 | 35
Amenorrhoea (Reproductive system and breast disorders) | 30 | 30
Genitourinary chlamydia infection (Infections and infestations) | 269 | 274
Urinary tract infection (Infections and infestations) | 223 | 281
Bacterial vaginosis (Infections and infestations) | 168 | 157
Vulvovaginitis trichomonal (Infections and infestations) | 149 | 158
Genitourinary tract gonococcal infection (Infections and infestations) | 143 | 160
Upper respiratory tract infection (Infections and infestations) | 140 | 139
Vulvovaginal candidiasis (Infections and infestations) | 148 | 127
Malaria (Infections and infestations) | 72 | 76
Gastroenteritis (Infections and infestations) | 61 | 59
Tonsillitis (Infections and infestations) | 54 | 57
Vaginal Infection (Infections and infestations) | 51 | 59
Vulvovaginitis (Infections and infestations) | 53 | 50
Respiratory tract infection (Infections and infestations) | 37 | 25
Folliculitis (Infections and infestations) | 29 | 26
Pelvic inflammatory disease (Infections and infestations) | 27 | 28
Alanine aminotransferase increased (Investigations) | 147 | 160
Aspartate aminotransferase increased (Investigations) | 144 | 145
Haemoglobin decreased (Investigations) | 125 | 143
Neutrophil count decreased (Investigations) | 118 | 146
Blood creatinine increased (Investigations) | 26 | 30
Abnormal loss of weight (Metabolism and nutrition disorders) | 173 | 175
Decreased appetite (Metabolism and nutrition disorders) | 25 | 26
Procedural pain (Injury, poisoning and procedural complications) | 79 | 95
Diarrhoea (Gastrointestinal disorders) | 30 | 39
Neutropenia (Blood and lymphatic system disorders) | 40 | 30
Anaemia (Blood and lymphatic system disorders) | 41 | 25
Headache (Nervous system disorders) | 41 | 45
Dysuria (Renal and urinary disorders) | 34 | 36

LIMITATIONS AND CAVEATS:
Dapivirine residual levels in used rings and dapivirine plasma concentrations are two objective measures of adherence to DVR ring use; however, they were found to be an imperfect measure of adherence as they cannot distinguish different patterns of use during the month. In addition, self-reported adherence based on the adherence questionnaires was also considered to have limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other